CLINICAL TRIAL: NCT04203680
Title: Efficacy of Histidine-Tryptophan-Ketoglutarate Solution Versus Blood Cardioplegia in Coronary Artery Bypass Graft Surgery: A Randomized Double Blinded Study
Brief Title: Histidine-Tryptophan-Ketoglutarate Solution Versus Blood Cardioplegia in CABG
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hoda Shokri, Assistant professor of Anaesthesiology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R 61/ 2019
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Cardioplegia Solution Adverse Reaction
MeSH Terms: interventions — Bretschneider cardioplegic solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HTK group (Sham Comparator): Patients received 30 ml/kg of HTK cardioplegic solution at 4°C through an antegrade fashion at an initial perfusion pressure of 80-100 mmHg
  Interventions: Drug: HTK cardioplegic solution
- blood cardioplegia group (Active Comparator): patients received one liter of blood cardioplegia was given with the antegrade route at 30°C, or lower. Blood maintenance cardioplegia was repeated every 30-45mins
  Interventions: Drug: blood cardioplegia

INTERVENTIONS:
Drug: HTK cardioplegic solution — 30 ml/kg of HTK cardioplegic solution at 4°C through an antegrade fashion at an initial perfusion pressure of 80-100 mmHg
  Other Names: Histidine-tryptophan-ketoglutarate solution
  Arms: HTK group
Drug: blood cardioplegia — one liter of blood cardioplegia was given with the antegrade route at 30°C, or lower. Blood maintenance cardioplegia was repeated every 30-45mins
  Arms: blood cardioplegia group

SUMMARY:
Background: In cardiac surgery, myocardial protection is mandatory during cross clamp time followed by reperfusion. Use of cardioplegic solutions preserves myocardial energy stores, hindering electrolyte disturbances and acidosis during periods of myocardial ischemia. This study was designed to compare the efficacy and safety of Histidine-tryptophan-ketoglutarate (HTK) solution versus blood cardioplegia in coronary artery bypass graft surgery.

Methods: Three hundred and twenty patients were randomized into Histidine-tryptophan-ketoglutarate (HTK) group and blood cardioplegia group. Ventilation time, total bypass time, cross clamp time, length of ICU or hospital stay and the early postoperative outcomes were analysed.

DETAILED DESCRIPTION:
The Ethics Committee of Ain Shams university approved this randomized prospective double-blinded controlled parallel group study to be held in Cardiothoracic Academy for three months from December 2019 to April 2020. The study was conducted on three hundred and twenty older patients aged from 60-80 years old posted for elective coronary artery bypass grafting (CABG). Written informed consents were signed by all patients. Exclusion criteria included (1) patients with Unstable angina (class III or IV); (2) Poor left ventricular function (LVEF <40%) ;(3) Patient with acute myocardial infarction; (4) Previous CABG; (5) Previous renal failure; (6) Preoperative Aortic valve or Mitral valve disease requiring replacement ;(7) Urgent CABG operation.

A detailed medical history, including medications used, symptoms and risk factors for ischemic heart disease (smoking, DM, hypertension), NYHA classification and full investigations were assessed on the night of the surgical procedure. Anesthesia management was standardized for all patients. Premedication with midazolam was limited to a maximum of 0.05 mg/kg. Anesthesia was done with 12 μg/kg fentanyl, 5-7 mg/kg thiopental sodium, and 0.15 mg/kg pancuronium and was maintained with 1-2.0% isoflurane. Heart rate and blood pressure were maintained within 20% of the baseline values. Anticoagulation was achieved with heparin 300 U/kg administered into the right atrium to maintain an activated clotting time above 480 s. Cardiopulmonary bypass (CPB) was established by non-occlusive roller pumps, membrane oxygenators and arterial line filtration. The CPB circuit was primed with 1.8 l lactated Ringer's solution and 50 ml of 20% mannitol. Management of CPB included systemic hypothermia during aortic cross-clamping, targeted mean perfusion pressure between 60 and 80 mmHg, and pump flow rates of 2.2 l/min/m2.Intraoperatively the patients were monitored using ECG, pulse oximetry, Invasive blood pressure monitoring, arterial blood gases, central venous line catheter and temperature probe. Surgical approach was performed by median sternotomy.

Patients were randomly allocated into 2 groups either HTK group and blood cardioplegia group according to a computer-generated randomization code, with allocation ratio 1:1. Opaque sealed envelopes were prepared according to the randomization schedule, and were opened by a clinician not involved in any part of the study.

In the HTK group, patients received 30 ml/kg of HTK cardioplegic solution at 4°C through an antegrade fashion at an initial perfusion pressure of 80-100 mmHg. In blood cardioplegia group, patients received one liter of blood cardioplegia was given with the antegrade route at 30°C, or lower. Blood maintenance cardioplegia was repeated every 30-45mins. The study medications were calculated and prepared by ICU residents who were not a part of the research team. To ensure blinding of study drug administration, the medication vials were kept in opaque bags. Trial bags were blinded and marked with a unique number. The allocation of trial drugs was determined by the web-based randomization system by the allocation of the bag number. The end-point assessor of the outcomes was blinded to the study drugs.

Before separation from CPB, patients were rewarmed to 36-37°C. After separation from CPB, heparin was neutralized with protamine sulfate 1 mg/100 U heparin to reach an activated clotting time within 10% of baseline. All patients were then transferred to the ICU after surgery.

The primary end-point of the study included early postoperative outcomes including cardiac enzymes preoperatively, 8 & 24 hour post-operatively, 30-day mortality, wall motion abnormalities and pericardial effusion. The secondary end-points included ventilation time, cross clamp and total bypass time, length of ICU stay, length of hospital stay, need for inotropic support, 30-day readmission, the incidence of late postoperative complications as renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* age from 60-80 years old
* elective CABG
* no comorbidities

Exclusion Criteria:

* patients with Unstable angina
* Poor left ventricular function
* Patient with acute myocardial infarction
* previous renal failure
* Preoperative Aortic valve or Mitral valve disease requiring replacement

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
mortality rate | up to 30 days postoperative
  mortality rate

SECONDARY OUTCOMES:
Troponin I level | Up to 24 hours postoperative
  level of troponin in the blood
length of ICU stay | up to 3 days postoperative
  ICU stay duration
length of hospital stay | up to 7 days postoperative
  hospital stay duration

CONTACTS AND LOCATIONS:
Overall Officials: Ayman shoeb, Study Chair — Ain Shams University
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 4 months
Access Criteria: Data were analyzed using SPSS Statistics version 23 (IBM© Corp., Armonk, NY, USA). Normally distributed numerical data were presented as mean and SD, and skewed data were presented as median and interquartile range. Qualitative data were presented as number and percentage or ratio. Normally distributed numerical data were compared using the unpaired t-test. Skewed numerical data were compared using the Mann-Whitney test and categorical data were compared using Fisher's exact test. P-value < 0.05 were considered statistically significant.